CLINICAL TRIAL: NCT00105066
Title: The Effects of Metformin on Vascular Structure and Function in Subjects With the Metabolic Syndrome (MET Trial)
Brief Title: The Effects of Metformin on Blood Vessel Structure and Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG0017
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Obesity; Hypertension; Hypercholesterolemia; Hyperglycemia
Keywords: Metabolic Syndrome; triglycerides; HDL; LDL; High Blood Pressure; High Cholesterol; High Blood Sugar
MeSH Terms: conditions — Obesity; Hypertension; Hypercholesterolemia; Hyperglycemia; Metabolic Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- Metformin (Experimental): Metformin 850 mg twice daily
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 850mg tablet once a day for one month, then twice a day for 3 months
  Other Names: Fortamet®; Glucophage®; Glumetza™; Riomet™
  Arms: Metformin
Drug: Placebo — placebo tablet once a day for one month, then twice a day for 3 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether the drug Metformin has beneficial effects on the blood vessels of individuals with the Metabolic Syndrome (MeS).

DETAILED DESCRIPTION:
Individuals with the Metabolic Syndrome (MeS) are at increased risk for developing cardiovascular diseases. This increased risk may, in part, be related to abnormalities in the blood vessels. MeS is defined as having 3 or more of the following 5 criteria:

* Abdominal obesity (waist measurement >39.8 inches in men, >34.4 inches in women)
* Elevated triglycerides (>150 mg/dl)
* Low HDL or "good" cholesterol (<40 mg/dl in men or <50 mg/dl in women)
* Elevated blood pressure (>130/85) or treatment for high blood pressure
* Elevated fasting blood sugar (>100 mg/dl)

Metformin is a medication that is approved by the Food and Drug Administration (FDA) for the treatment of diabetes; however, it can also be safely administered to non-diabetic subjects. We are evaluating whether Metformin reduces the stiffness of blood vessels and improves endothelial function.

This study requires 4 visits to the NIA Clinical Research Center (located on the premises of Harbor Hospital) over a 5-month period. At the initial visit, patients will be given a physical examination with blood and urine tests, and an EKG. They will be randomized into one of two groups; one group will receive Metformin (1700 mg per day), while the other group will receive a placebo. Participants will take the medication for 4 months. Subsequent visits will include additional blood tests, ultrasound and echo exams.

Taking part in this study is entirely voluntary. All testing and medications will be provided at no cost to the participant or their family.

ELIGIBILITY:
Inclusion Criteria:

Participants with the Metabolic Syndrome, which is defined as having 3 or more of the following 5 alterations:

* Abdominal obesity (waist measurement >39.8 inches in men, >34.4 inches in women)
* Elevated triglycerides (>150 mg/dl)
* Low HDL or "good" cholesterol (<40 mg/dl in men or <50 mg/dl in women)
* Elevated blood pressure (>130/85) or treatment for high blood pressure
* Elevated fasting blood sugar (>100 mg/dl)

Exclusion Criteria:

* Diabetes treated with medication
* Blood pressure >160/100 mmHg
* Clinical Congestive Heart Failure
* Anemia with hematocrit <32%
* Asthma or Chronic Obstructive Pulmonary Disease (COPD) requiring daily medication or use of home oxygen therapy
* Major surgery planned within the next six months
* A recent, unexplained weight loss of >10% of body weight in the past 6 months
* A known allergy or hypersensitivity to Metformin
* History of hepatitis or cirrhosis
* History of kidney disease (defined as serum creatinine >1.4 mg/dL in men, >1.3 mg/dL in women)
* Pregnancy or the absence of an effective method of contraception
* Illicit drug or alcohol abuse
* Cancer requiring treatment currently or recently completed treatment in the last 2 months

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2004-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Ferrucci, MD, Principal Investigator — National Institute on Aging (NIA); James Strait, M.D., Ph.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute on Aging (NIA), Harbor Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Beisswenger PJ, Howell SK, Touchette AD, Lal S, Szwergold BS. Metformin reduces systemic methylglyoxal levels in type 2 diabetes. Diabetes. 1999 Jan;48(1):198-202. doi: 10.2337/diabetes.48.1.198. PMID 9892243
- [Background] Mather KJ, Verma S, Anderson TJ. Improved endothelial function with metformin in type 2 diabetes mellitus. J Am Coll Cardiol. 2001 Apr;37(5):1344-50. doi: 10.1016/s0735-1097(01)01129-9. PMID 11300445
- [Background] Effect of intensive blood-glucose control with metformin on complications in overweight patients with type 2 diabetes (UKPDS 34). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):854-65. PMID 9742977

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo : placebo tablet once a day for one month, then twice a day for 3 months
- Metformin: Metformin : 850mg tablet once a day for one month, then twice a day for 3 months
Period: Overall Study
Arm/Group | Placebo | Metformin
Started | 27 | 50
Completed | 25 | 45
Not Completed | 2 | 5
Not completed — Adverse Event | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Metformin | Total
Number analyzed (Participants) | 27 | 49 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (13.5) | 55.1 (11.8) | 54.4 (12.7)
Gender [Count of Participants; unit: Participants]
  Female | 19 | 34 | 53
  Male | 8 | 15 | 23
Carotid Femoral Pulse Wave Velocity [Mean (Standard Deviation); unit: meters/second] | 6.8 (2.1) | 6.8 (2.1) | 6.8 (2.1)
FMD [Mean (Standard Deviation); unit: percentage] — Flow Mediated Dilation of brachial artery (percent change in blood flow after hyperemia)
  percentage | 7.6 (4.4) | 9.3 (6.1) | 8.5 (5.3)
HOMA-S [Mean (Standard Deviation); unit: HOMA Score] — HOMA Insulin Sensitivity Index
  HOMA Score | 52.9 (26.9) | 52.3 (23.1) | 52.5 (24.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Arterial Stiffness Compared to Baseline
Time Frame: Baseline and 4.5 months
Measure: Mean (Standard Deviation); unit: meters / second
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 25 | 45
meters / second | -7.2 (2.1) | -7.3 (1.8)

2. Primary Outcome: Change in Flow Mediated Dilation (FMD)
Description: to evaluate improvement in endothelial function
Time Frame: Baseline and 4.5 months
Population: Participants with complete data.
Measure: Mean (Standard Deviation); unit: percentage change in diameter
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 23 | 39
percentage change in diameter | 8.8 (7.0) | 10.5 (8.0)

3. Post Hoc Outcome: Homa Insulin Sensitivity
Description: Homeostatic Model Assessment of insulin sensitivity
Time Frame: 4.5 months
Population: Participants with complete data.
Measure: Mean (Standard Deviation); unit: HOMA Score
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 23 | 39
HOMA Score | 57.4 (36.3) | 64.5 (27.7)

ADVERSE EVENTS:
Arm/Group | Placebo | Metformin
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/50
Other Adverse Events (participants affected / at risk) | 1/27 | 6/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Metformin (N=50)
Nausea (Gastrointestinal disorders) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No